CLINICAL TRIAL: NCT05183061
Title: Factors Associated With Post-induction Hypotension in Idiopathic Normal Pressure Hydrocephalus (iNPH) Patient Undergoing Ventriculoperitoneal (VP) and Lumbar Peritoneal (LP) Shunt
Brief Title: Factors Associated With Post-induction Hypotension in iNPH Patient Undergoing VP and LP Shunt
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phuriphong Songarj, Associate Professor, Mahidol University
Other Study IDs: 961/2563(IRB4)
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: The iNPH Patients Scheduled for VP or LP Shunt Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypotensive group: Hypotenson is defined as systolic blood pressure (SBP) < 80 mmHg or a drop more than 20% from baseline SBP for longer than 10 minutes or a drop that requires treatment either vasopressor or inotropic drugs.
  Interventions: Drug: Ehedrine Norepineprine
- Non-hypotensive group: The pateints who did not develop hypotensive episodes as aforementioned.

INTERVENTIONS:
Drug: Ehedrine Norepineprine — No interventions required considering that this was a retrospective study.
  Groups: Hypotensive group

SUMMARY:
This study is a retrospective work involving the review of patients who were scheduled for VP or LP shunt in Siriraj Hospital, Mahidol University, Thailand. The sample size calculation was based on the rule of thumbs of the logistic regression comprising 18 risk factors. The incidence of post-induction hypotension according to our institution's pilot study November 2019-January 2020) was 47%. With 10% addition for missing data and other possible reasons, the sample size was 426. The primary objective of the study is to report the factors associated with post-induction hypotension in iNPH patients undergoing VP or LP shunt procedures. Our secondary objective is to determine the incidence of post-induction hypotension in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective cases of iNPH scheduled for VP and LP shunt
* Patients aged > 18 years old

Exclusion Criteria:

* Emergency cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Elective cases of iNPH scheduled for VP and LP shunt whose medical records were acquired from the hospital's central database.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Factors associated with post-induction hypotension in iNPH patients undergoing VP or LP shunt procedures | 9 months
  Risk factors associated with post-induction hypotension after administration of anesthetic agents

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology Department, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No